CLINICAL TRIAL: NCT05409586
Title: Evaluating the Risk Factors and the Role of Albumin-to-globulin Ratio in Predicting Recurrence Among Patients With Idiopathic Granulomatous Mastitis
Brief Title: Risk Factors and the Role of Albumin-to-globulin Ratio in Idiopathic Granulomatous Mastitis
Status: Completed | Type: Observational
Sponsor: Samsun Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Ahmet Burak Ciftci, Director, Samsun Education and Research Hospital
Other Study IDs: SAMSUNERH.IGM
Record Dates: First submitted 2022-05-29; First posted 2022-06-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Idiopathic Granulomatous Mastitis
Keywords: Idiopathic granulomatous mastitis; recurrence; albumin-to-globulin ratio; risk factors
MeSH Terms: conditions — Recurrence | interventions — Mastectomy, Segmental; Drainage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- no recurrence: Patients who recovered after IGM treatment and had no signs of relapse
  Interventions: Procedure: segmental mastectomy
- recurrence: Patients whose symptoms reappear 3 months after IGM treatment
  Interventions: Procedure: segmental mastectomy

INTERVENTIONS:
Procedure: segmental mastectomy — The preferred method in the treatment of some patients diagnosed with IGM
  Other Names: Incision and Drainage

SUMMARY:
Albumin-to-globulin ratio (AGR) is an inflammation-based index that has been shown to have a role in many cancers and inflammatory diseases. Idiopathic granulomatous mastitis (IGM) is a rare inflammatory disease of the breast with a high recurrence rate. As a relatively new biomarker for inflammatory diseases, AGR's role in IGM recurrence has never been investigated in the literature. This study primarily investigates the possible risk factors for IGM recurrence and whether AGR can be used as a predictive factor.

DETAILED DESCRIPTION:
Patients diagnosed with IGM on pathology reports between January 2016 and March 2021 were enrolled in the study and their medical records were analyzed retrospectively. The patients were divided into two groups: recurrence and non-recurrence. Clinical, demographic characteristics, and laboratory parameters were compared. The best cut-off value for significant factors in predicting recurrence was determined by receiver operating characteristic (ROC) analysis. Univariate and multivariate logistic regression analysis was used to determine the risk factors that are effective in IGM recurrence.

ELIGIBILITY:
Inclusion Criteria:

* The patients with a pathologically confirmed diagnosis of granulomatous mastitis
* Patients over the age of 18
* Female patients

Exclusion Criteria:

* Male patients
* Secondary granulomatous mastitis etiologies (tuberculous mastitis and Wegener's granulomatosis)
* Patients who do not have enough follow-up information
* Patients with missing data

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with IGM on pathology reports between January 2016 and March 2021
Sampling Method: Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-05-25 (Actual)

PRIMARY OUTCOMES:
IGM recurrence | within an average of 3-4 years of follow-up after treatment
  Recurrence was defined as the reappearance of breast complaints such as pain, mass, abscess, and fistula at the end of at least three months following remission with treatment. IGM developed in the other breast after the treatment was also accepted as a recurrent case.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsun Eğitim ve Araştırma Hastanesi, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The datasets generated and analyzed in this study will be available from the corresponding author on reasonable request.

REFERENCES:
- [Background] Xuan Q, Yang Y, Ji H, Tang S, Zhao J, Shao J, Wang J. Combination of the preoperative albumin to globulin ratio and neutrophil to lymphocyte ratio as a novel prognostic factor in patients with triple negative breast cancer. Cancer Manag Res. 2019 May 31;11:5125-5131. doi: 10.2147/CMAR.S195324. eCollection 2019. PMID 31213922
- [Result] Uysal E, Soran A, Sezgin E; Granulomatous Mastitis Study Group. Factors related to recurrence of idiopathic granulomatous mastitis: what do we learn from a multicentre study? ANZ J Surg. 2018 Jun;88(6):635-639. doi: 10.1111/ans.14115. Epub 2017 Jul 27. PMID 28749045
- [Result] Azizi A, Prasath V, Canner J, Gharib M, Sadat Fattahi A, Naser Forghani M, Sajjadi S, Farhadi E, Vasigh M, Kaviani A, Omranipour R, Habibi M. Idiopathic granulomatous mastitis: Management and predictors of recurrence in 474 patients. Breast J. 2020 Jul;26(7):1358-1362. doi: 10.1111/tbj.13822. Epub 2020 Apr 5. PMID 32249491
- [Result] Velidedeoglu M, Kundaktepe BP, Aksan H, Uzun H. Preoperative Fibrinogen and Hematological Indexes in the Differential Diagnosis of Idiopathic Granulomatous Mastitis and Breast Cancer. Medicina (Kaunas). 2021 Jul 8;57(7):698. doi: 10.3390/medicina57070698. PMID 34356979
- [Derived] Ciftci AB, Buk OF, Yemez K, Polat S, Yazicioglu IM. Risk Factors and the Role of the Albumin-to-Globulin Ratio in Predicting Recurrence Among Patients with Idiopathic Granulomatous Mastitis. J Inflamm Res. 2022 Sep 18;15:5401-5412. doi: 10.2147/JIR.S377804. eCollection 2022. PMID 36158516